

Abbreviation: IIF: Individual Information Form; OKT: Osteoporosis Knowledge Test; OHBS: Osteoporosis Health Belief Scale; OSES: Osteoporosis Self-Effective Scale; IPAQ: International Physical Activity Questionnaire Short Form; IMB Model: Information- Motivation and Behavior Skills Model.

## **Study Protocol**